CLINICAL TRIAL: NCT01431196
Title: Phase II Trial With Autologous Dendritic Cell Vaccination in Patients With Stage II-III HER2 Negative Breast Cancer
Brief Title: Trial With Autologous Dendritic Cell Vaccination in Patients With Stage II-III HER2 Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Marta Santisteban, MD, PhD, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEND/CM
Record Dates: First submitted 2011-04-01; First posted 2011-09-09 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Stage II Breast Cancer; Stage III Breast Cancer
Keywords: breast cancer; neoadjuvant chemotherapy; autologous dendritic cell vaccination
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DENDRITIC CELL VACCINATION (Experimental): Px will receive standard neoadjuvant chemotherapy plus active vaccination. we will compare results with an historic cohort of patients treated with the same chemotherapy without the vaccines
  Interventions: Biological: Autologous dendritic cell vaccination

INTERVENTIONS:
Biological: Autologous dendritic cell vaccination — Autologous dendritic cell vaccination. Dendritic cells are pulsed with their own tumor antigens

SUMMARY:
Molecular expression in breast cancer (BC) defines special fenotypes with different prognostic and predictive features.Since the addition of trastuzumab and lapatinib to chemotherapy, HER2 overexpressing tumors have become the best responders to systemic therapies, reaching pathologic complete response rates (pCR) around 50%. But HER2 negative tumors (luminal A and triple negative) are characterized by low chemosensitivity (luminal A) or early distant relapse after diagnosis (triple negative BC) . In this open, prospective, non-randomized and multicentric phase II study the investigators include stage II and III HER2 negative BC patients that are going to receive neoadjuvant sequential chemotherapy Epirubicin+Ciclofosfamide x 4 and then Docetaxel x 4)with an individualized vaccination with autologous dendritic cells pulsed with their own tumor. The hypothesis is that the reinforcement of the immune system with the autologous dendritic cell vaccination against HER2 negative BC could increase pathologic complete responses (pCR) and disease free survival(DFS), when added to chemo, surgery and radiation therapy and in a maintenance schedule.

DETAILED DESCRIPTION:
Chemotherapy schedule:

* dose dense epirubucin 100 mgr/m2 plus ciclofosfamide 600 mgr/m2 every two weeks for four cycles with with GM-CSF support on day +1 (pegylated filgastrim) or on days +5 to +9 (filgastrim) subcutaneously
* docetaxel 80-100 mgr/m2 every three weeks for four cycles. Addition of GM-CSF if docetaxel doses are > 85 mgr/m2

ELIGIBILITY:
Inclusion Criteria:

* HER2 negative and stage II and III Breast cancer patients who benefit with neoadjuvant chemotherapy
* age 18-75
* to get enough tumoral sample to elaborate the vaccine

Exclusion Criteria:

* pregnancy
* severe diseases
* hepatitis or HIV
* need to be on immunosuppressant drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
pathologic complete response (pCR) in the breast and the axilla | 6 months after starting chemotherapy

SECONDARY OUTCOMES:
Number of participants with adverse events | During the 6-24 months of administration of the vaccine
Impact of the vaccine on patients DFS and OS | three to five years after the diagnosis of breast cancer
  We will compare our cohort of patients vaccinated and treated with chemotherapy, surgery and radiation therapy with an historic cohort in our center treated with the same schedule of chemotherapy , surgery and radiation therapy without the vaccine
EORTC quality of life | From 9 months and up to two years
Correlation among the specific immune response induced in patients and the pathologic response of the tumor | 6-24 months
  Specific immune response will be evaluated as delayed hipesrsensitivity (DTH), humoral response by cuantification antibodies against tumoral cells (ELISA)and cellullar response (proliferation assay and citokines production)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Santisteban, MD, PhD., Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clínica Universidad de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
By 2017 scientific data should be communicated

REFERENCES:
- [Derived] Santisteban M, Solans BP, Hato L, Urrizola A, Mejias LD, Salgado E, Sanchez-Bayona R, Toledo E, Rodriguez-Spiteri N, Olartecoechea B, Idoate MA, Lopez-Diaz de Cerio A, Inoges S. Final results regarding the addition of dendritic cell vaccines to neoadjuvant chemotherapy in early HER2-negative breast cancer patients: clinical and translational analysis. Ther Adv Med Oncol. 2021 Dec 23;13:17588359211064653. doi: 10.1177/17588359211064653. eCollection 2021. PMID 34987618